CLINICAL TRIAL: NCT05666713
Title: NHLBI Transmural Electrosurgery LeafLet Traversal and Laceration Evaluation (TELLTALE) BASILICA-TAVR Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10000673; 000673-H
Record Dates: First submitted 2022-12-24; First posted 2022-12-28 (Actual); Results first posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Valvular Heart Disease; Aortic Valve Failure
Keywords: Structural heart disease interventions; TAVR; TAVR Associated Coronary Artery Obstruction; Electrosurgery; Native Aortic Valve Failure; Bioprosthetic Aortic Valve Failure
MeSH Terms: conditions — Heart Valve Diseases; Hyperthermia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Participants undergoing TAVR with BASILICA using Transmural TELLTALE guidewire system (Experimental): Participants with severe aortic stenosis or failure of surgically-implanted bioprosthetic valve undergoing transcatheter aortic valve replacement (TAVR) with bioprosthetic or native aortic scallop intentional laceration to prevent iatrogenic coronary artery obstruction (BASILICA) using the Transmural TELLTALE guidewire system.
  Interventions: Device: TELLTALE BASILICA procedure

INTERVENTIONS:
Device: TELLTALE BASILICA procedure — The TELLTALE BASILICA procedure has five steps: (1) engagement of the target leaflet with a guiding catheter; (2) electrosurgical leaflet traversal with the TELLTALE guidewire, (3) preparation and positioning of the TELLTALE guidewire electrosurgical leaflet laceration surface; (4) electrosurgical leaflet laceration with the TELLTALE guidewire, immediately followed by (5) TAVR. These are all guided by fluoroscopy, with adjunctive echocardiography as needed.
  Other Names: Transmural TELLTALE guidewire system

SUMMARY:
Background:

Replacing a valve in the heart can save many people's lives. The procedure is called transcatheter aortic valve replacement (TAVR). In rare cases, a flap of tissue called a leaflet can shift during TAVR; the leaflet may block blood flow to the coronary arteries, which supply blood to the heart muscle. About 50% of people who experience this problem will die. To reduce this risk, doctors will cut this leaflet during TAVR. But the tools used to cut the leaflet were originally designed for other purposes. Using these tools during TAVR can be complicated and risky. Researchers want to make TAVR safer.

Objective:

To test a new device (TELLTALE) designed specifically for use during TAVR.

Eligibility:

People aged 21 years and older who are undergoing TAVR and who are at high risk of coronary artery obstruction.

Design:

Participants will be screened. They will have routine tests that are done before undergoing TAVR.

Before the procedure, participants will complete a questionnaire. They will talk about how their heart disease affects their quality of life. Their physical abilities and their risk of stroke will be assessed.

Participants will be admitted to the hospital for TAVR. They will be placed under general anesthesia or moderate sedation. The procedure will be performed using the TELLTALE guidewire system.

Participants will repeat the tests of their physical abilities after the procedure. They will also repeat the questionnaire about their quality of life. These will be repeated again at a follow-up visit in 30 days.

Participants will have a final study visit after 90 days. This visit may be in person or remote.

DETAILED DESCRIPTION:
Transcatheter aortic valve implantation (TAVR) may cause life threatening coronary artery obstruction, whether implanted in native aortic stenosis or bioprosthetic aortic valve failure.

We have developed and validated the techniques of BASILICA (Bioprosthetic Aortic Scallop Intentional Laceration to prevent Iatrogenic Coronary Artery obstruction during transcatheter aortic valve replacement), using bedside modification of off-the-shelf guidewires. These bedside modifications require additional assembly steps and special expertise, and thereby risks procedure failure and complications.

Transmural Systems and NHLBI have developed a purpose-built electrosurgical guidewire system (TELLTALE) to simplify the BASILICA-TAVR procedure. The purpose of this protocol is to test the efficacy and safety of this purpose-built guidewire in the setting of BASILICA-TAVR.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in the study, candidates must meet all of the following criteria:

* Adults age >= 21 years
* High or prohibitive risk of surgical aortic valve replacement according to the local multidisciplinary heart team
* Undergoing TAVR for bioprosthetic aortic valve failure or native aortic stenosis ( on-label TAVR)
* Local multidisciplinary heart team determines subject to be at high risk of TAVR-induced coronary artery obstruction
* Deemed likely to suffer coronary artery obstruction from TAVR based on NHLBI Core lab analysis of CT, any of

  * Risk is narrow Sinus of Valsalva: (a) Leaflet height is greater than coronary artery height, and (b) Virtual transcatheter valve-to-coronary (VTC) distance < 4mm
  * Risk is Sinus sequestration: (a) Threatening leaflet height is greater than sinotubular junction, and (b) Virtual transcatheter valve-to-sinotubular-junction distance (VTS) < 2mm at the affected Sinus
* Concurrence of the Study Eligibility Committee
* Able to understand the protocol, consents in writing to participate, and willing to comply with all study procedures for the duration of the study

EXCLUSION CRITERIA:

* Requires doppio (two-leaflet) BASILICA
* Flail target leaflet at baseline
* Excessive target aortic leaflet calcification (no basal calcium-free window or potentially obstructive calcific masses) on baseline CT
* Planned provisional (pre-position coronary artery) stents despite BASILICA
* Requires non-femoral access
* Requires concomitant procedures during TAVR (such as percutaneous coronary intervention for baseline obstructive coronary artery disease)
* Chronic kidney disease KDIGO stage 4 or 5 (eGFR < 29 ml/min/1.73m2) or renal replacement therapy
* Not expected to survive for 12 months
* Pregnant at the time of intended treatment (day 0)

Ages: 21 Years to 109 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-02-21 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2025-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Lederman, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (10):
- United States (10):
  - California Pacific Med Ctr, San Francisco, California
  - University of Colorado Health, Fort Collins, Colorado
  - Medstar WHC, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Rochester Regional Health, Rochester, New York
  - St. Francis Hospital and Heart Center, Roslyn, New York
  - Montefiore Medical Center, The Bronx, New York
  - Carilion Medical Center, Roanoke, Virginia
  - University of Washington Heart Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant results data will be made available 6 months after publication date for a period of 5 year by sending a request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be made available 6 months after publication date for a period of 5 year
Access Criteria: Sending request to Robert.Lederman@nih.gov

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Participants Undergoing TAVR With BASILICA Using Transmural TELLTALE Guidewire System
Started | 90
Completed | 89
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Participants Undergoing TAVR With BASILICA Using Transmural TELLTALE Guidewire System
Number analyzed (Participants) | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 85
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59
  Male | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 81
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 82
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 90

OUTCOME MEASURES:

1. Primary Outcome: Number of Participant That Experienced Technical Success With the TELLTALE Guidewire System
Description: The primary efficacy endpoint is technical success, which is defined when the following criteria are all met:
  1. Successful electrosurgical leaflet traversal using the TELLTALE Guidewire
  2. Successful electrosurgical leaflet laceration using the TELLTALE Guidewire
  3. Successful retrieval of the TELLTALE Guidewire System
Time Frame: 1 minute following procedure discharge (Exit from the catheterization laboratory)
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Undergoing TAVR With BASILICA Using Transmural TELLTALE Guidewire System
Number analyzed (Participants) | 90
Participants | 90

2. Primary Outcome: Number of Inpatient Safety Events
Description: Inpatient safety as defined by:
  1. Freedom from all-cause mortality as defined as the total number of deaths from any cause
  2. Freedom from stroke, both disabling and non-disabling
     * Disabling stroke according to VARC-3 is defined as a stroke resulting in significant, persistent neurological deficits that impact a patient's ability to perform daily activities.
     * Non-disabling stroke according to VARC-3, involves stroke symptoms that don't significantly impair a patient's ability to perform daily activities or lead to a worsening of their pre-stroke disability level.
  3. Freedom from acute coronary artery obstruction
  4. Freedom from emergency cardiac surgery or reintervention related to the TELLTALE BASILICA procedure or device-
  5. Freedom from BASILICA-related complications including coronary artery perforation, coronary artery dissection, aortic dissection, cardiac free wall perforation, or systemic embolization of a native or bioprosthetic leaflet
Time Frame: Upon discharge from the index hospital admission, up to 30 days
Measure: Number; unit: Safety Events
Arm/Group | Participants Undergoing TAVR With BASILICA Using Transmural TELLTALE Guidewire System
Number analyzed (Participants) | 90
Safety Events
  All-cause Mortality | 0
  Stroke, disabling | 1
  Stroke, non-disabling | 2
  Coronary obstruction | 1
  Emergency cardiac surgery or reintervention | 0
  BASILICA related complications | 0

3. Secondary Outcome: Freedom From Safety Events
Description: 30-day safety as assessed by freedom from
  * Major Adverse Cardiovascular Events defined by no periprocedural myocardial infarction, cerebrovascular events, and periprocedural all-cause mortality
  * All-cause mortality: defined as total number of deaths from any cause
  * All stroke (disabling and non-disabling per VARC-3)
    * Disabling results in significant, persistent neurological deficits that impact daily activities
    * Non-disabling involves stroke symptoms that don't significantly impair daily activities or lead to worsening of their pre-stroke level
  * Bleeding VARC-3 Type 2 or greater requiring two or more units of transfused blood or hemoglobin drop >3g/dL
  * Major vascular, access-related, or cardiac structural complication according to VARC-3, including coronary obstruction
  * Acute kidney injury stage 3 or 4
  * Moderate or severe aortic regurgitation
  * New permanent pacemaker due to procedure-related conduction abnormalities
  * Surgery or intervention related to the TELLTALE device
Time Frame: Up to Day 30
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants Undergoing TAVR With BASILICA Using Transmural TELLTALE Guidewire System
Number analyzed (Participants) | 90
percentage of participants | 89 [80 to 94]

ADVERSE EVENTS:
Time Frame: Up to 90 Days
Description: All adverse events (AE) and adverse device effects (ADE) through the 30 days follow-up will be reported. All serious adverse device effects (SADE), serious adverse events (SAE), unanticipated device effects (UADE), and unanticipated problems (UP) will be recorded through the 90 days follow up.
Arm/Group | Participants Undergoing TAVR With BASILICA Using Transmural TELLTALE Guidewire System
All-Cause Mortality (participants affected / at risk) | 0/90
Serious Adverse Events (participants affected / at risk) | 36/90
Other Adverse Events (participants affected / at risk) | 62/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Undergoing TAVR With BASILICA Using Transmural TELLTALE Guidewire System (N=90)
Bronchial Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 8 (8)
Heparin Induced Thrombocytopenia (HIT) (Blood and lymphatic system disorders) | 1 (1)
Arterial injury (Injury, poisoning and procedural complications) | 5 (5)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Acute coronary obstruction post TAVR (Injury, poisoning and procedural complications) | 1 (1)
Injury to jugular vein (Injury, poisoning and procedural complications) | 2 (2)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Arterial thromboembolism (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Thromboembolic event (Vascular disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Atrioventricular block complete (Cardiac disorders) | 5 (5)
Conduction disorder (Cardiac disorders) | 1 (1)
Heart failure (Cardiac disorders) | 3 (6)
Sick sinus syndrome (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Creatinine increased (Investigations) | 2 (2)
Delirium (Psychiatric disorders) | 1 (1)
Endocarditis infective (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Skin infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (2)
Urinary retention (Renal and urinary disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Reoccurrence of Mantle Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1)
Stroke (Nervous system disorders) | 6 (7)
Total right hip arthroplasty (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Undergoing TAVR With BASILICA Using Transmural TELLTALE Guidewire System (N=90)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Creatinine increased (Investigations) | 8 (9)
Cardiac troponin I increased (Investigations) | 19 (19)
Ejection fraction decreased (Investigations) | 1 (1)
TELLTALE guidewire Non-target traversal (Investigations) | 6 (6)
Platelet count decreased (Investigations) | 9 (9)
Anemia (Blood and lymphatic system disorders) | 15 (15)
Hematocrit decreased post procedure (Blood and lymphatic system disorders) | 1 (1)
B-cell lymphoma (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 8 (8)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1)
Arterial thromboembolism (Injury, poisoning and procedural complications) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Coccyx pain (Injury, poisoning and procedural complications) | 1 (1)
Minor Groin bleed (Injury, poisoning and procedural complications) | 11 (11)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 6 (6)
Cardiac troponin I increased (Cardiac disorders) | 19 (19)
Chest pain - cardiac (Cardiac disorders) | 5 (5)
Conduction disorder (Cardiac disorders) | 16 (17)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Fever (General disorders) | 3 (3)
Non-cardiac chest pain (General disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Memory impairment (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Trigeminal nerve disorder (Nervous system disorders) | 1 (1)
Hematoma (Vascular disorders) | 3 (3)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 6 (6)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Scrotal infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (4)
Urinary retention (Renal and urinary disorders) | 3 (3)
Mobitz (type) II atrioventricular block (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-10-31): https://cdn.clinicaltrials.gov/large-docs/13/NCT05666713/Prot_SAP_001.pdf
  • Informed Consent Form (2024-11-01): https://cdn.clinicaltrials.gov/large-docs/13/NCT05666713/ICF_000.pdf